CLINICAL TRIAL: NCT03477045
Title: Can Oils Derived From Genetically-modified Plants Replace Fish Oil as a Source of Long Chain n-3 Polyunsaturated Fatty Acids in the Human Diet
Brief Title: Does Consuming Modified Plant Seed Oil Containing Fish Oil Fatty Acids Act in the Same Way as Consuming Fish Oil?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 17497
Record Dates: First submitted 2018-03-07; First posted 2018-03-26 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Healthy
Keywords: omega 3 polyunsaturated fatty acid; camelina sativa; fatty acid composition; immune modulation
MeSH Terms: interventions — Fish Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fish oil (Active Comparator): Fish oil providing 450 mg of eicosapentaenoic acid plus docosahexaenoic acid per dose
  Interventions: Dietary Supplement: Single dose fish oil; Dietary Supplement: single dose Camelina seed oil
- Camelina seed oil (Experimental): Camelina seed oil providing 450 mg of eicosapentaenoic acid plus docosahexaenoic acid per dose
  Interventions: Dietary Supplement: Repeated dose fish oil; Dietary Supplement: repeated dose camelina seed oil

INTERVENTIONS:
Dietary Supplement: Single dose fish oil — Fish oil consumed within a single high fat test meal
  Arms: Fish oil
Dietary Supplement: Repeated dose fish oil — Fish oil consumed daily for 8 weeks
  Arms: Camelina seed oil
Dietary Supplement: single dose Camelina seed oil — camelina seed oil consumed within a single high fat test meal
  Arms: Fish oil
Dietary Supplement: repeated dose camelina seed oil — camelina seed oil consumed daily for 8 weeks
  Arms: Camelina seed oil

SUMMARY:
Fish oil and oily fish contain omega 3 long chain polyunsaturated fatty acids known to be beneficial to health. Many people consume little, despite UK government recommendations to eat at least one portion of oily fish per week. Furthermore, despite modest consumption, fish stocks are declining due to over fishing. Therefore, there is a need for an alternative, sustainable and cost efficiently produced dietary source. A seed oil source of these fish oil-type fatty acids has been achieved by adding genes from other plant sources to the oil seed plant Camelina sativa. Camelina sativa, related to mustard and cabbage, has provided seed oil for human consumption for thousands of years. It was the most important oil seed plant in Europe until the 1900's. This research is being done to see if consuming fish oil-type fatty acids in Camelina seed oil allows the body to take up and use the fish oil fatty acids in the same way as it does from fish oil.

DETAILED DESCRIPTION:
This research is being done to see if consuming fish oil-type omega 3 long chain polyunsaturated fatty acids in Camelina seed oil allows the body to take up the fish oil fatty acids in the same way as it does from fish oil.

In the first study (A) the Camelina oil will be used in a meal. The volunteers (healthy men and women) will be asked to consume the meal and provide blood samples in the following 6 hours to look at immediate uptake of the fish oil fatty acids. This will be repeated (for comparison) with fish oil.

The second study (B) will look at consumption over a longer period. Volunteers will be asked to consume the Camelina oil daily for 8 weeks and provide blood samples at the visits at the start and end of that period. This will be repeated (for comparison) with fish oil.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. 18 to 30 years or 50 to 65 years
3. Body mass index 18.5-30.0 kg/m2
4. Health screening results that are within normal clinical ranges
5. Not consuming fish oil or other oil supplements
6. Not eating more than one oily fish meal per week
7. Willing to adhere to the study protocol
8. Being able to provide written informed consent

Exclusion Criteria:

1. Aged < 18 years; 31-49 years or > 65 years
2. Body mass index < 18.5 or > 30 kg/m2
3. Current smoker
4. Fasting blood cholesterol or glucose concentrations outside the normal concentration range
5. Diagnosed chronic illness (for example diagnosed cardiovascular disease, diabetes, cancer)
6. Use of prescribed medicine to control inflammation
7. Use of prescribed medication to control blood lipids (e.g. statins, fibrates (fenofibrate), Omacor)
8. Use of prescribed medication to control blood pressure (ACE inhibitors, angiotensin 2 receptor blockers, calcium channel blockers, α-inhibitors, thiazide diuretics)
9. Use of fish oil or other oil supplements
10. Chronic gastrointestinal problems (e.g. IBD, coeliac disease, cancer)
11. Pregnant or planning to become pregnant within the study period
12. Participation in another clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2019-11-04 (Actual)

PRIMARY OUTCOMES:
Uptake of omega 3 polyunsaturated fatty acids after short term consumption of fish oil or Camelina seed oil. | Short term consumption - single dose followed over 8 hours
  The magnitude of the increase in omega 3 polyunsaturated fatty acids in plasma lipids and blood cells following consumption of modified Camelina seed oil for short (postprandial) period compared with fish oil.
Uptake of omega 3 polyunsaturated fatty acids after longer term consumption of fish oil or Camelina seed oil. | Longer term consumption daily for 8 weeks. Follow up at 8 weeks.
  The magnitude of the increase in omega 3 polyunsaturated fatty acids in plasma lipids and blood cells following consumption of modified Camelina seed oil for 8 weeks compared with fish oil.

SECONDARY OUTCOMES:
Effect of omega 3 polyunsaturated fatty acid consumption on postprandial inflammatory markers after consumption of fish oil or Camelina seed oil. | Short term consumption - single dose followed over 8 hours
  To measure the appearance of inflammatory mediators in the blood of healthy subjects over 8 hours following consumption of a standard high fat meal containing modified Camelina seed oil compared with consuming the same meal containing fish oil.
Effect of omega 3 polyunsaturated fatty acid consumption for 8 weeks on in vitro immune responses after consumption of fish oil or Camelina seed oil. | Longer term consumption daily for 8 weeks. Follow up at 8 weeks.
  To measure in vitro immune responses (immune cells inflammatory markers and response to bacterial challenge) by peripheral blood mononuclear cells following consumption of modified Camelina seed oil for 8 weeks compared with consuming fish oil for the same duration.

CONTACTS AND LOCATIONS:
Overall Officials: Graham C Burdge, PhD, Principal Investigator — University of Southampton
Locations (1):
- Faculty of Medicine, University of Southampton, Southampton, Hants, United Kingdom

REFERENCES:
- [Result] West AL, Michaelson LV, Miles EA, Haslam RP, Lillycrop KA, Georgescu R, Han L, Sayanova O, Napier JA, Calder PC, Burdge GC. Differential postprandial incorporation of 20:5n-3 and 22:6n-3 into individual plasma triacylglycerol and phosphatidylcholine molecular species in humans. Biochim Biophys Acta Mol Cell Biol Lipids. 2020 Aug;1865(8):158710. doi: 10.1016/j.bbalip.2020.158710. Epub 2020 Apr 11. PMID 32289503
- [Result] West AL, Miles EA, Lillycrop KA, Han L, Napier JA, Calder PC, Burdge GC. Dietary supplementation with seed oil from transgenic Camelina sativa induces similar increments in plasma and erythrocyte DHA and EPA to fish oil in healthy humans. Br J Nutr. 2020 Nov 14;124(9):922-930. doi: 10.1017/S0007114520002044. Epub 2020 Jun 9. PMID 32513312
- [Result] West AL, Michaelson LV, Miles EA, Haslam RP, Lillycrop KA, Georgescu R, Han L, Napier JA, Calder PC, Burdge GC. Lipidomic Analysis of Plasma from Healthy Men and Women Shows Phospholipid Class and Molecular Species Differences between Sexes. Lipids. 2021 Mar;56(2):229-242. doi: 10.1002/lipd.12293. Epub 2020 Dec 7. PMID 33284478
- [Result] West AL, Miles EA, Lillycrop KA, Napier JA, Calder PC, Burdge GC. Genetically modified plants are an alternative to oily fish for providing n-3 polyunsaturated fatty acids in the human diet: A summary of the findings of a Biotechnology and Biological Sciences Research Council funded project. Nutr Bull. 2021 Mar;46(1):60-68. doi: 10.1111/nbu.12478. Epub 2020 Dec 23. PMID 33776584

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-18): https://cdn.clinicaltrials.gov/large-docs/45/NCT03477045/Prot_SAP_000.pdf